CLINICAL TRIAL: NCT07153198
Title: Promoting Socioemotional Development in Early Childhood: Implementation and Evaluation of the VIPP-SD Parenting Intervention in Portugal
Acronym: SAF-Parents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida (Other)
Responsible Party: Principal Investigator, Maria Manuela Pedro Veríssimo, Professor, ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: I-011-04-25; Grant nº 325160 (Other Grant/Funding Number: Calouste Gulbenkian Foundation)
Record Dates: First submitted 2025-07-05; First posted 2025-09-03 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-08

CONDITIONS: Parent-Child Relations
Keywords: sensitivity; attachment; behavioral problems; economic advantages
MeSH Terms: conditions — Hypersensitivity; Problem Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with VIPP-SD (Active Comparator): Intervention group:
  Interventions: Other: VIPP-SD
- Control Group: No intervention (No Intervention): No Intervention

INTERVENTIONS:
Other: VIPP-SD — Consists of four sessions (with the option of one or two additional booster sessions), held biweekly, depending on the family's needs and availability. Specifically, VIPP-SD addresses disciplinary strategies alongside sensitivity themes through: (1) the differentiation between attachment and exploration behaviors; interpretation of child's behavior and significance of a sensitive response to it; and the importance of sharing emotions (2) the application of distraction and induction as non-coercive techniques in response to challenging child behaviours or conflict-prone situations; (3) the utilization of positive reinforcement, whereby parents praise adaptive behaviours and ignore maladaptive, attention-seeking actions; (4) the implementat of a sensitive interaction pause to de-escalate conflict or temper tantrums; and (5) the demonstration of empathy towards the child in conjunction with consistent disciplinary approaches and explicit boundary-setting
  Arms: Intervention with VIPP-SD

SUMMARY:
The Video-feedback Intervention to Promote Positive Parenting and Sensitive Discipline (VIPP-SD) is an attachment-based intervention aimed at promoting parental sensitivity and the use of developmentally appropriate, non-coercive discipline strategies (ref). The VIPP-SD intervention integrates the enhancement of parental sensitive responsiveness (Ainsworth et al., 1974) with parent coaching aimed at preventing coercive parent-child interaction cycles (Patterson, 1982) and facilitating sensitive limit-setting practices.ase parental sensitivity and sensitive discipline of the primary parent

DETAILED DESCRIPTION:
Aims and hypotheses

1. The primary aim of the Growing Minds - Strengthening Affective Bonds is to demonstrate the effect of the VIPP-SD on parental sensitivity and sensitive discipline of the primary parent, 8 weeks after the intervention and six months after the intervention. It is expected that sensitivity and sensitive discipline of parents in the intervention condition will significantly increase post-intervention, compared to sensitivity and sensitive discipline of parents in the control condition, who have a similar number of ('dummy') contacts with the interveners.
2. The secondary aim of the study is to examine the efficacy of the intervention in reducing children's behavioral problems, as a function of increased parental sensitivity and the use of sensitive discipline strategies. It is expected that improvements in parenting behaviors resulting from the VIPP-SD intervention will be associated with lower levels of behavioral difficulties in children over time.
3. A third objective of the study is to evaluate the impact of the intervention on broader parenting practices and parental well-being, specifically aiming to mitigate psychopathological symptomatology. The focus will be on reducing symptoms of depression and anxiety among participating parents, in line with evidence suggesting that improvements in parenting sensitivity may contribute to enhanced parental mental health.
4. Finally, the investigators will examine whether the intervention yields economic advantages for society at large. To do this, the investigators will use quality-adjusted life-years (QALYs) as the unit of outcome, allowing to quantify health benefits. By comparing the QALYs associated with the intervention to those resulting from no intervention, the investigators aim to assess the cost-effectiveness and potential return on investment from a societal perspective. This analysis will help determine whether the intervention not only improves family relations but also contributes to economic efficiency by potentially reducing healthcare costs, improving productivity, and enhancing overall societal well-being

ELIGIBILITY:
Inclusion Criteria: Children will be between 2 and 6 years old, and their parents between must be fluent in Portuguese -

Exclusion Criteria: Children with disabilities, chronic illnesses, or hereditary diseases will be excluded from the study

-

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Parental sensitivity: Erickson Scales of Parental Sensitivity (ESPS, Egeland, et al., 1990) | Data will be collected at pretest, posttest (14 weeks) .
  Parental sensitivity will be assessed using the the revised Erickson 7-point rating scales for Supportive Presence (from 1 = parent completely fails to be supportive to the child to 7 = parent skilfully provides support throughout the session) and Intrusiveness (from 1 = parent allows the child sufficient time to explore and to attempt to solve tools on her/his own to 7 = parent is highly intrusive; her agenda clearly has precedence over the child's wishes; Egeland et al., 1990). Supportive presence is defined as the consistent emotional, physical, and psychological availability of a mother, characterized by both verbal expressions and nonverbal behaviors. High sensitivity is associated with positive developmental outcomes in children, including secure attachment and better emotional regulation. Intrusiveness reflects the extent to which a parent disregards or interferes with the child's autonomy, wishes, interests, or behaviors.

SECONDARY OUTCOMES:
Strengths & Difficulties Questionnaire" (SDQ Portuguese version Fleitlich et al., 2004) | Data will be collected at pretest, posttest (14 weeks) and follow up (12 weeks).
  The assessment tool used in this study is a 25-item questionnaire designed to evaluate emotional and behavioral problems in children aged 2 to 17 years, with responses provided by parents. The items are rated on a 3-point scale: 0 = "Not true," 1 = "A bit true," and 2 = "Very true." The questionnaire is structured into five subscales: (1) emotional symptoms, (2) conduct problems, (3) hyperactivity, (4) peer problems, and (5) prosocial behavior. For this study, only the parent version of the questionnaire is utilized. The total difficulties score is derived by summing the first four subscales (excluding prosocial behavior), yielding a score ranging from 0 to 40.
Depression, Anxiety, and Stress Scale - 21 (DASS-21) | Data will be collected at pretest, posttest (14 weeks) and follow up (12 weeks).
  The Depression, Anxiety, and Stress Scale - 21 (DASS-21; Lovibond & Lovibond, 1995; Portuguese version: Apóstolo et al., 2006) is a 21-item self-report questionnaire designed to assess symptoms of depression, anxiety, and stress in parents. Each item is rated on a 4-point Likert scale ranging from 0 (Did not apply to me at all) to 3 (Applied to me most of the time). The scale comprises three subscales: Depression (7 items), which assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest or involvement, anhedonia, and inertia; Anxiety (7 items), which measures autonomic arousal, skeletal muscle effects, situational anxiety, and the subjective experience of anxious affect; Stress (7 items), which evaluates chronic, nonspecific arousal, including difficulty relaxing, nervous arousal, irritability, agitation, and impatience. Subscale and total scores are calculated by summing the item responses.
AQOL-8D (Richardson & Lezzi, 2014) | Data will be collected at pretest, posttest (14 weeks) and follow up (12 weeks).
  Quality of life among caregivers will be measured with the Assessing Quality of Life - 8 Dimensions (AQOL-8D) (Richardson & Lezzi, 2014) is a multi-attribute utility instrument developed to provide a sensitive and comprehensive assessment of health status among adults across eight dimensions,, including independent living, mental health, coping, relationships, pain, self-worth, happiness and senses) and 35 items with four to six response levels, each representing increasing levels of severity. This measure will be used for economic evaluation.
Resource Use Characterization Questionnaire. | Data will be collected at pretest, posttest (14 weeks) and follow up (12 weeks).
  Resources used by children and their parents will be measured using a questionnaire adapted from published questionnaires by Bouwmans et al, 2013 and Pokhilenko et al. 2023. Resource use will include healthcare services (accident and emergency visits, primary care and specialized outpatient visits and inpatient stays, medication), social services, transportation, absenteeism and presenteeism from both paid and unpaid work, and out-of-pocket expenses. This measure will be used for economic evaluation.
Child Rearing Practices Report-Questionnaire (CRPR-Q) | Data will be collected at pretest, posttest (14 weeks) and follow up (12 weeks).
  The Child Rearing Practices Report-Questionnaire (CRPR-Q; Rickel & Biasatti, 1982, Ribeiro et al, 2021) is a 40-item parent-report questionnaire used to assess parenting practices that are theoretically and empirically linked to child developmental outcomes. Parents are instructed to respond with reference to a specific child in the household, rating each item on a 6-point Likert scale ranging from 1 (strongly disagree) to 6 (strongly agree). The measure comprises two theoretically grounded subscales: Nurturance and Restrictiveness

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Verissimo, PhD, Principal Investigator — ISPA - Instituto Universitario de Ciencias Psicologicas, Sociais e da Vida
Locations (1):
- Manuela Verissimo, Lisbon, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No
Intellectual Property Data (IPD) might not be shared due to concerns about confidentiality and legal restrictions. Sharing it could risk exposing proprietary or sensitive information, including details that may affect entire family's privacy.

REFERENCES:
- [Derived] Verissimo M, Guedes M, Fernandes M, Fernandes C, Santos C, Diniz E, Oliveira P, Negrao M, Sampaio F, Bakermans-Kranenburg M. Promoting socioemotional development in early childhood: implementation and evaluation of the VIPP-SD parenting intervention in Portugal. BMC Psychol. 2025 Oct 29;13(1):1190. doi: 10.1186/s40359-025-03431-3. PMID 41163103